CLINICAL TRIAL: NCT00854503
Title: Metabolic and Vascular Effects of Statins in Untreated Dyslipidemic Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Davide Lauro, University of Rome Tor Vergata
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 131/08
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-01

CONDITIONS: Type 2 Diabetes; Diabetic Dyslipidemia
Keywords: Statins administration in diabetic dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Simvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Simvastatin (Active Comparator): Simvastatin 20 mg/day
  Interventions: Drug: Simvastatin
- Rosuvastatin (Active Comparator): Rosuvastatin 20 mg/day
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Simvastatin — 20 mg/day in one oral administration
  Arms: Simvastatin
Drug: Rosuvastatin — 20 mg/day in one oral administration.
  Arms: Rosuvastatin

SUMMARY:
Type 2 diabetes (T2D), because of impaired glucose regulation and consequent hyperglycemia, promotes the development of coronary heart disease. Secondary dyslipidemia is often associated with T2D and enhances the risk of cardiovascular complications. HMG-CoA reductase inhibitors (statins) are selectively administrated for the treatment of dyslipidemia, leading to a significant reduction of cardiovascular risk. More recently, revisions to guidelines have established a lower therapeutic LDL cholesterol goal for diabetic patients, requiring the administration of higher dose of statin. However, it is unclear whether high dose statin therapy could affect glycemic control in diabetic patients. Moreover, data regarding the effects of statins on insulin-resistance and endothelial function are controversial.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes in good glycemic control, treated with metformin alone.
* Untreated dyslipidemia.
* BMI <30.

Exclusion Criteria:

* History of cancer.
* History of cardiovascular diseases.
* Any other acute or cronic illness which requires administration of steroids or other drugs able to interfere with glucose metabolism.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance assessed by HbA1c and fasting glucose | 1, 6, 12 months

SECONDARY OUTCOMES:
insulin-resistance assessed by clamp. Endothelial function assessed by FMD %. Inflammatory status assessed by biochemical markers. | 1, 6, 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rome Tor Vergata, Rome, Italy